CLINICAL TRIAL: NCT06164899
Title: Long-term Evaluation of Outcomes of Patients Undergoing Autologous Bone Marrow Concentrate Infiltration vs. Hyaluronic Acid for the Treatment of Bilateral Knee Osteoarthritis. Prospective Observational Study
Brief Title: Long-term Evaluation of Outcomes of Patients Undergoing Autologous Bone Marrow Concentrate Infiltration vs. Hyaluronic Acid
Status: Completed | Type: Observational
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Other Study IDs: OA-bi Blind LT
Record Dates: First submitted 2023-12-01; First posted 2023-12-11 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Knee Osteoarthritis
Keywords: hyaluronic acid injection; BMAC injection; Bone Marrow aspirate concentrate; long term follow-up; Prospective observational study; Hyalorunic acid; knee joint
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with bilateral knee osteoarthritis treated with hyaluronic acid injection: Patients with bilateral osteoarthritis treated with hyaluronic acid injection treated within the research protocol "OA-bi-blind"
- Patients with bilateral knee osteoarthritis treated with BMAC injection: Patients with bilateral knee osteoarthritis treated with autologous bone marrow concentrate injection treated within the research protocol "OA-bi-blind"

SUMMARY:
This is a prospective observational study for long-term clinical evaluation (minimum 4-year follow-up) in patients treated within the research protocol "OA-bi-blind" (Double-blind randomized trial on the treatment of bilateral knee osteoarthritis: Autologous bone marrow concentrate VS. hyaluronic acid)

DETAILED DESCRIPTION:
60 patients treated within the "OA-bi-blind" research protocol from 2016 to 2019 at the II Orthopaedic and Trauma Clinic of the Rizzoli Orthopaedic Institute will be recruited. These are patients undergoing infiltration for the treatment of bilateral gonarthrosis of autologous bone marrow concentrate vs. hyaluronic acid within the OA-bi-Blind Research protocol.Prior to enrollment, patients will be contacted provided they have released their personal or legal guardian's e-mail address and/or personal or legal guardian's telephone number in advance and only after verifying the patient's consent to be contacted again for research purposes. If the patient is interested in participating in the study, arrangements will be made with him or her to send the Informed Consent and Disclosure Letter.

The patient will have to return (by means of a pre-stamped envelope that he will have received together with the consent itself) the Informed Consent completed in all its parts to the address given in the information letter. Only upon obtaining the fully completed Informed Consent may the investigator subject the patient to a telephone interview.

Alternatively, the patient may receive the Informed Consent and the questionnaire for clinical evaluations digitally.Clinical score data will be collected from the questionnaires conducted at long-term follow-up of patients enrolled in the study. The data collected during the long-term follow-up, will be used to evaluate the time course of outcomes after treatment with autologous bone marrow concentrate versus hyaluronic acid in patients who received either treatment as per the ''OA-bi-blind'' protocol.

ELIGIBILITY:
Inclusion Criteria:

-Patients undergoing injection for the treatment of bilateral gonarthrosis of autologous bone marrow concentrate vs. hyaluronic acid within the OA-bi-Blind Research protocol at the II Orthopedic and Trauma Clinic of the Rizzoli Orthopedic Institute.

Who met the following criteria at the time of treatment:

* Male or female patients, aged 18 to 75 years;
* Symptomatic bilateral knee osteoarthritis (Kellgren-Lawrence grade 1-4);
* Failure after at least 2 months of conservative treatment;
* Ability and consent of patients to actively participate in the rehabilitation protocol and clinic and radiological follow-up; And who meet the following criteria at the time of assessment by telephone or via telemedicine platform;
* Capable patients
* Signature of informed consent
* Availability

Exclusion Criteria:

* Patients no longer on call;
* Patients who do not agree to undergo evaluation
* Patients who have passed away.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing infiltration for the treatment of bilateral gonarthrosis of autologous bone marrow concentrate vs. hyaluronic acid within the OA-bi-Blind Research Protocol at the II Orthopedic and Trauma Clinic of the Rizzoli Orthopedic Institute
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2024-02-09 (Actual); Primary Completion 2025-02-12 (Actual); Study Completion 2025-02-12 (Actual)

PRIMARY OUTCOMES:
Knee Injury and Osteoarthritis Outcome Score (IKDC)-Subjective Knee Evaluation Form | baseline
  This is a subjective, knee-specific rating scale that is considered one of the most reliable assessment tools in the evaluation of knee pathology. The questionnaire examines 3 categories: symptoms, sports activity, and knee function. According to this questionnaire, a score between 0 and 100 can be obtained, where a high score is associated with a high level of function and minor pain symptoms. A score of 100 is in fact interpreted as a condition in which there are neither limitations in conducting activities of daily living nor symptoms.
Knee Injury and Osteoarthritis Outcome score- (KOOS Score) | baseline
  The full questionnaire consists of five subscales and they cover: pain (9 items), symptoms (7 items of which two relate to stiffness), functions and activities of daily living (17 items) physical function, sports activities and leisure (5 items) and quality of life in relation to the knee (4 items). All items in the relevant subscales have the same response mode, use a 5-point Likert scale, and each question is assigned a score from 0 to 4, where 0 indicates "no difficulty" and 4 "a severe difficulty). Score range 0-100 for each subscale
EuroQol Visual Analogue Scale (EQ-VAS ) | baseline
  This is a visual analog scale that has a range of scores from 0 (worst imaginable health condition) to 100 (best imaginable health condition).
Tegner Score | baseline
  This questionnaire allows the estimation of a subject's motor activity level with a score between 0 and 10, where 0 represents 'inability' and 10 represents 'participation in competitive sports, such as soccer at the national or international level. This score is the one most commonly used to define the motor activity level of patients with knee disorders. In the study, the Tegner Score will be filled in directly by the investigator, through an interview the patient. In addition, questions will also be asked about return to sports and pre-injury, pre-treatment and recovered/achieved sports level .
EQ-5D (EuroQoL) Current Health Assessment | baseline
  EQ-5D is a standardized measure of health-related quality of life developed by the EuroQol Group to provide a simple generic questionnaire for use in clinical and economic evaluation and population health surveys
Patient Acceptable Symptom State (PASS) | baseline
  A tool to assess patient satisfaction in consideration of their current degree of pain, function, and daily activity. Patients can express if their state of health will be satisfying, answering "yes" or "no.
Visual Analogue Scale (VAS) | baseline
  Visual analog scale consisting of a straight line segment (10 cm length), the ends of which correspond to "no pain" (0) and "the strongest pain imaginable" (10).
Final treatment opinion | baseline
  The patient should indicate satisfaction and relative degree with the treatment performed after a minimum of 4 years after infiltrative treatment. All patients will be able to indicate their health condition by choosing from this answers: much better", "somewhat better", "no change", "a little worse", "much worse".
Failure | baseline
  The patient will be asked to indicate whether and when new infiltrative or surgical treatment was performed. Questions will also be asked about any complications and reinterventions

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Zaffagnini, MD, Principal Investigator — Istituto Ortopedico Rizzoli - II Clinica Ortopedica e Traumatologica
Locations (1):
- Istituto Ortopedico Rizzoli, Bologna, Italy

REFERENCES:
- [Background] Boffa A, Di Martino A, Andriolo L, De Filippis R, Poggi A, Kon E, Zaffagnini S, Filardo G. Bone marrow aspirate concentrate injections provide similar results versus viscosupplementation up to 24 months of follow-up in patients with symptomatic knee osteoarthritis. A randomized controlled trial. Knee Surg Sports Traumatol Arthrosc. 2022 Dec;30(12):3958-3967. doi: 10.1007/s00167-021-06793-4. Epub 2021 Nov 12. PMID 34767030
- [Background] Cavallo C, Boffa A, Andriolo L, Silva S, Grigolo B, Zaffagnini S, Filardo G. Bone marrow concentrate injections for the treatment of osteoarthritis: evidence from preclinical findings to the clinical application. Int Orthop. 2021 Feb;45(2):525-538. doi: 10.1007/s00264-020-04703-w. Epub 2020 Jul 13. PMID 32661635
- [Background] Filardo G, Madry H, Jelic M, Roffi A, Cucchiarini M, Kon E. Mesenchymal stem cells for the treatment of cartilage lesions: from preclinical findings to clinical application in orthopaedics. Knee Surg Sports Traumatol Arthrosc. 2013 Aug;21(8):1717-29. doi: 10.1007/s00167-012-2329-3. Epub 2013 Jan 11. PMID 23306713
- [Background] Fortier LA, Strauss EJ, Shepard DO, Becktell L, Kennedy JG. Biological Effects of Bone Marrow Concentrate in Knee Pathologies. J Knee Surg. 2019 Jan;32(1):2-8. doi: 10.1055/s-0038-1676069. Epub 2018 Nov 30. PMID 30500973
- [Background] Trigkilidas D, Anand A. The effectiveness of hyaluronic acid intra-articular injections in managing osteoarthritic knee pain. Ann R Coll Surg Engl. 2013 Nov;95(8):545-51. doi: 10.1308/rcsann.2013.95.8.545. PMID 24165334